CLINICAL TRIAL: NCT05383924
Title: Patient's Compliance to Intrauterine Device: Immediate Postplacental Insertion Versus Delayed Insertion in Women Undergoing Planned Cesarean Section
Brief Title: Intrauterine Contraceptive Device Insertion During Cesarean Section (CS) Versus Delayed Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Rania Hassan Mostafa, Principal investigator, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FMASU MS720/2021
Record Dates: First submitted 2022-05-14; First posted 2022-05-20 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Contraception; IUD
Keywords: IUD; immediate postplacental IUD; interval IUD insertion; compliance; expulsion
MeSH Terms: conditions — Patient Compliance

STUDY DESIGN:
Intervention Model Description: This study aims to compare immediate postplacental IUD insertion versus delayed insertion as regards patient's compliance in women undergoing planned cesarean section. One group will have the IUD inserted during cesarean section. Another group will undergo IUD insertion after 6 weeks of delivery by CS.
Masking Description: masking is not applicable
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postplacental IUD (PP-IUD) insertion (Active Comparator): patients will have immediate postplacental IUD insertion
  Interventions: Procedure: postplacental IUD insertion
- delayed IUD insertion (Active Comparator): cesarean section will be done, then contacts will be taken to arrange for delayed IUD insertion at the 6th week postpartum visit
  Interventions: Procedure: delayed IUD insertion

INTERVENTIONS:
Procedure: postplacental IUD insertion — patients will have immediate postplacental IUD insertion as follows: The IUD is inserted after removal of the placenta and after the uterus has become hemostatic. After initiating closure of the uterine incision, the IUD is placed at the top of uterine fundus manually. Before closing the uterine incision, the strings are placed gently in the lower uterine segment manually. After this is accomplished, the uterine incision closure can be completed. The strings will usually descend spontaneously through the cervix during the puerperal period. If the cervix is closed, it'll be dilated from above with ring forceps. Strings can be passed through the cervix with ring forceps. If this is done, the surgeon will recheck to make sure IUD remains at the fundus of the uterus prior to closing the uterine incision. Strings can be trimmed at a follow-up visit.
  Ultrasound will be done after the CS to ensure proper placement of the IUD.
  Other Names: immediate postplacental IUD insertion
  Arms: postplacental IUD (PP-IUD) insertion
Procedure: delayed IUD insertion — cesarean section will be done, then contacts will be taken to arrange for delayed IUD insertion at the 6th week postpartum visit as follows: Prepare IUD prior to starting procedure Place vaginal speculum then prepare vaginal wall with betadine Apply tenaculum at anterior cervical position then insert and remove uterine sound Place IUD according to package insert then cut threads 2-3 cm from cervical os. Ultrasound will be done to ensure proper placement of the IUD.
  Other Names: interval IUD insertion
  Arms: delayed IUD insertion

SUMMARY:
After ethical committee approval and written consent from the patients, this prospective quasi-randomized controlled clinical trial was performed on pregnant women planning to deliver by cesarean section and willing to participate in the study to investigate the value of immediate post placental IUD insertion versus delayed insertion on patient's compliance in Ain Shams University Maternity Hospital (ASUMH).

DETAILED DESCRIPTION:
* After protocol approval by the ethical committee of the department of Obstetrics & Gynecology, Faculty of Medicine, Ain Shams University; pregnant woman planning to undergo elective cesarean section in ASUMH were recruited from the antenatal clinic.
* Counselling was done about different postpartum contraceptive methods including immediate PPIUD and delayed IUD insertion.
* An informed written consent was taken from all participants before enrollment in the study and after explaining the purpose, possible risks and complications.
* History taking, examination, and investigations (CBC, follow-up Ultrasound) were done to identify eligible patients according to the inclusion and exclusion criteria.
* Randomization: Eligible patients were quasi-randomized into 2 groups:

Group (A) (PPIUD group): immediate postplacental IUD insertion. Group (B) (delayed insertion group): delayed IUD insertion at the 6th week postpartum visit.

Randomization was done through "Alternation" method.

- Allocation: the first patient (no.1) was allocated to group (A) and second patient (no.2) to group (B) and so on by ''Alternation method '' till fulfilling the sample size.

Procedure:

Type of IUD: Model T-shaped Copper 380 A: Safe-load® or Pregna®

* Group A (PPIUD group): cesarean section (CS) was performed by experts in post-placental IUD insertion as follows: The IUD was inserted after removal of the placenta and after the uterus had become hemostatic. After initiating closure of the uterine incision, the IUD was placed at the top of uterine fundus manually. Before closing the uterine incision, the strings were placed gently in the lower uterine segment manually. After this was accomplished, the uterine incision closure could be completed. The strings usually descended spontaneously through the cervix during the puerperal period. If the cervix was closed, it would be dilated from above with ring forceps. Strings can be passed through the cervix with ring forceps. If this was done, the surgeon would recheck to make sure IUD remains at the fundus of the uterus prior to closing the uterine incision. Strings can be trimmed at a follow-up visit. Ultrasound was done after the CS to ensure proper placement of the IUD.
* Group B (control group) (delayed insertion group): cesarean section was done by expert supervisors, then contacts were taken to arrange for delayed IUD Insertion at the 6th week postpartum visit as follows: IUD was prepared prior to starting procedure. Vaginal speculum was placed then prepared vaginal wall with betadine. Tenaculum was applied at anterior cervical position then uterine sounding was performed. IUD was placed according to package insert, then the threads were cut 2-3 cm from cervical os. Ultrasound was done to ensure proper placement of the IUD.
* Follow-up: follow-up visits were conducted at 6, 12months post-insertion (questionnaire, ultrasound, hemoglobin level).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women planned for delivery by cesarean section in Ain Shams University Maternity hospital

Exclusion Criteria:

* Women not consenting to use IUD as a contraceptive method and preferring other methods.
* Any woman with condition included in Category 3 or 4 for Cu-IUD in medical eligibility criteria for contraceptive use World Health Organization (WHO) 2015
* Neuropsychiatric disorder causing altered mentality or perception
* Intrapartum complications as chorioamnionitis, massive blood loss, or hysterectomy.
* Anemic patients (hemoglobin level <10g/dl).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
Patient compliance | at 6 months after the procedure
  compliance to IUD will be assessed by a user satisfaction questionnaire with scoring system: Q1, on a scale from 0 to 10, Are You satisfied of using Cu-IUD as a contraceptive method? (When 0 means "Not at all satisfied" and 10 means "Extremely Satisfied") 0 1 2 3 4 5 6 7 8 9 10 Q2, Will you continue to use Cu-IUD in future or reuse it after discontinuation? 1 = Yes 0 = No Q3, Do you recommend Cu-IUD for others to use it as a contraceptive method?
  1 = Yes 0 = No
Patient compliance | at 12 months after the procedure
  compliance to IUD will be assessed by a user satisfaction questionnaire with scoring system: Q1, on a scale from 0 to 10, Are You satisfied of using Cu-IUD as a contraceptive method? (When 0 means "Not at all satisfied" and 10 means "Extremely Satisfied") 0 1 2 3 4 5 6 7 8 9 10 Q2, Will you continue to use Cu-IUD in future or reuse it after discontinuation? 1 = Yes 0 = No Q3, Do you recommend Cu-IUD for others to use it as a contraceptive method?
  1 = Yes 0 = No

SECONDARY OUTCOMES:
Abnormal Bleeding pattern | at 12 months after the procedure
  heavy menstrual bleeding or other abnormal uterine bleeding as reported by history taking
dyspareunia | at 12months after the procedure
  pain during intercourse, as reported by history taking
Efficiency | at 6 months after the procedure
  successful insertion and proper position of the IUD, as confirmed by ultrasound imaging
Efficiency | at 12 months after the procedure
  proper position of the IUD, as confirmed by ultrasound imaging
Anemia | at 12months after the procedure
  hemoglobin drop by follow-up of hemoglobin level after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Sweed, MD, Study Chair — Faculty of Medicine Ain Shams University
Locations (1):
- Ain Shams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
upon reasonable request to the principal investigator, individual participant data can be shared
Supporting Information: Study Protocol, Analytic Code
Time Frame: individual participant data with supporting information will be available after study completion for 6 months after publication
Access Criteria: reasonable requests aiming for extending the benefit to more patients, or asking about the procedures done, will be assessed by the principal investigator and/or the study official, and shared either by contact e-mails or data repository when available